CLINICAL TRIAL: NCT02444481
Title: Open Multicenter Clinical Study of the Efficacy of the Local Treatment With Polygynax of Mycotic and/or Bacterial Vaginitis
Brief Title: Open Study of the Efficacy of the Local Treatment With Polygynax of Bacterial and/or Mycotic Vaginitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoire Innotech International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGX401-08
Record Dates: First submitted 2013-05-14; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Vaginitis
Keywords: Mycotic Vaginitis
MeSH Terms: conditions — Vaginitis | interventions — Neomycin; Nystatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polygynax, antibiotic, vaginal treatment (Experimental): Polygynax combinaison of nystatine, polymyxin, neomycin, Local treatment of vaginal infection during 12 days. One vaginal capsule every evening.
  Interventions: Drug: Polygynax combinaison of polymyxin, Neomycin and Nystatin

INTERVENTIONS:
Drug: Polygynax combinaison of polymyxin, Neomycin and Nystatin

SUMMARY:
Open prospective multicenter phase IV study in patients presenting with symptoms of bacterial and/or mycotic (mushroom) vaginitis for 12 days as specified in the product information.

Investigators/centers: 20 gynacologists are previewed to do the study in ambulatory treatment.

Objectifs of the study:

Principal objectif:

Evaluation of the efficacy of the treatment on the clinical symptoms of bacterial and/or mycotic vaginitis

Secondary objectif:

Evaluation of the efficacy of the treatment on eradication of the diagnosed germs Evaluation of the correspondence of the efficacy on the symptoms and on the eradication of the germs.

Numbers of patients previewed: 100 patients for evaluation of the efficacy

Criteria of evaluation

Principal criteria:

Clinical efficacy as judged by the investigator Secondary criteria:evaluation of clinical symptoms judged by the patient reduction or emlimination of bacteria and other germs the relationship between clinical and bacterial results

Evaluation of tolerance

Used Study Drug:

Polygynax, vaginal capsule consisting of Polymyxin 35000 UI, Neomycin 35000UI and Nystatin 100000UI Application: vaginal application once daily in the evening for 12 days

Study design:

Visit 1:

All patients presenting with the clinical symptoms, presenting all inclusion criteria and none of the exclusion criteria are included in the study at visit 1 and receive Polygynax treatment (one vaginal capsule once daily in the evening).

A vaginal smear is obtained. Visit 2 (optional) If the results of the bacteriological examination confirms an infection with germs sensible to the treatment with Polygynax the treatment is continued. If other germs not sensible to Polygynax are present, the patients is contacted to stop the treatment, to come back to a second visit to her gynacologist who will change the treatment. The other patients continue the treatment.

Visit 3:

After the treatment the patients come back to the last visit. A clinical evaluation and a vaginal smear for control is obtained.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 years to 65 years
* Agreeing to provide written informed consent
* Presenting symptoms of vaginitis: unaccustomed leucorrhoea, pruritus, burning sensation on micturition, dyspareunia.

Exclusion Criteria:

* Patients in menstrual period,
* Virgins,
* Clinically detectable sexually transmissible infections (STI): genital lesions, evocative leucorrhoea, recent history of STI (< 3 months), known STI in partner,
* Sexually transmissible disease, including HIV,
* Pregnancy,
* Breastfeeding,
* Known allergy or hypersensitivity to the treatment or to any of the ingredients of the treatment, and in particular, hypersensitivity to soya oil,
* Use of male or female condoms,
* Use of spermicide,
* Use of diaphragm,
* Clinical symptoms of non-sensitive bacterial vaginosis: runny and unpleasant smelling leucorrhoea suggesting Gardnerella vaginalis vaginitis,
* Concomitant topical or systemic anti-infective treatment,
* Topical or systemic anti-infective treatment in the 14 days prior to the study,
* Immunodepression or any other major disease rendering completion of the study or interpretation of the study results difficult,
* Immunosuppressant therapy,
* Chemotherapy,
* Participation in another clinical trial in the month prior to the study,

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy on clinical symptoms as judged by the investigator | 14 days
  Clinical efficacy is judged upon symptoms

SECONDARY OUTCOMES:
Bacteriological efficacy on reduction of the presence of bacteria and /or fungus | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Bohbot, Principal Investigator — Institut Alfred Fournier